CLINICAL TRIAL: NCT00633841
Title: Randomized, Controlled, Parallel Group, Patient-Blinded, Single-Center Phase I Pilot Study to Assess Tolerability and Safety of Repeated s.c. Administration of a Single-Dose of AFFITOPE AD02 Applied With or Without Adjuvant to Patients With Mild to Moderate Alzheimer's Disease
Brief Title: Tolerability and Safety of Subcutaneous Administration of AFFITOPE AD02 in Mild to Moderate Alzheimer's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Affiris AG (Industry)
Responsible Party: Affiris GmbH
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Affiris 002
Record Dates: First submitted 2008-03-05; First posted 2008-03-12 (Estimated); Last update posted 2010-10-19 (Estimated); Status verified 2010-10

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer; Morbus Alzheimer; Alzheimer Vaccine; Vaccine; AD; Aβ immunotherapy
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): AFFITOPE AD02 without adjuvant
  Interventions: Biological: AFFITOPE AD02
- 2 (Active Comparator): AFFITOPE AD02 with adjuvant
  Interventions: Biological: AFFITOPE AD02

INTERVENTIONS:
Biological: AFFITOPE AD02 — 4 subcutaneous injections of IP in 4-week intervals

SUMMARY:
The purpose of this study is to assess the tolerability and safety of repeated subcutaneous injection of a single dose of AFFITOPE AD02 in patients with mild to moderate Alzheimer's Disease.

DETAILED DESCRIPTION:
Alzheimer's Disease (AD) is a devastating neurodegenerative disorder for which there is no cure.

Although the etiology of AD is not fully understood, recent research suggests that Aβ is central to the disease process. Consequently, approaches capable of removing Aβ from the brain, such as Aβ immunotherapy, are expected to possess disease-modifying potential. This view is supported by evidence gathered in mouse models of AD and studies involving AD patients.

Based on the view that active Aβ immunotherapy has disease-modifying potential both in animal models of AD and in patients, and on the knowledge gathered on the side-effects of Aβ-based immunotherapy encountered in humans, we designed a new generation of AD vaccines. Rather than using full length Aβ itself, we choose to use mimotopes of the N-terminal end of Aβ as the antigenic component of our vaccine (Mimotopes discovered by Affiris GmbH have been termed AFFITOPES). Mimotopes are peptides that functionally mimic the native antigenic epitope but do not show sequence identity to it. Thus, while being different from the original antigen, mimotopes are recognized by the same antibodies and, vice versa, are capable of inducing antibodies that cross-react with the original antigen itself. A major advantage offered by mimotopes is the lack of tolerance mechanisms that would prevent the induction of an immune response to it (as is the case with self peptides/proteins such as Aβ). To further increase the vaccine's safety profile, the length of the mimotope used was limited to preclude the elicitation of Aβ-specific T cells. Also, the mimotope used has been designed to generate antibodies directed exclusively to Aβ (i.e., they do not recognize parental APP itself). To provide helper epitopes for the generation of an antibody response, the mimotope is coupled to a carrier.

The trial is designed as a patient-blinded, single-center, randomized, controlled, parallel group, phase I clinical study of repeated once every 4 weeks administration by subcutaneous injection of AFFITOPE AD02 alone or adsorbed to aluminium hydroxide in 24 patients with mild to moderate Alzheimer's Disease. In total, each patient will receive 4 immunizations. Patients will be randomized to receive AFFITOPE AD02 alone or adsorbed to alumimium hydroxide. Each treatment group consists of 12 patients. For safety reasons, inclusion of patients will be done in a stepwise manner.

ELIGIBILITY:
Main Inclusion Criteria:

* Diagnosis of probable Alzheimer's disease based on the NINCDS/ADRDA criteria.
* Alzheimer's disease of mild to moderate degree (MMSE 16-26)
* Magnetic Resonance Imaging scan (MRI) of brain consistent with diagnosis of AD.
* Written informed consent signed and dated by the patient and the caregiver.
* Age 50-80 years.
* Availability of a partner/caregiver

Other Inclusion Criteria apply.

Main Exclusion Criteria:

* Presence or history of allergy to components of the vaccine.
* Contraindication for MRI imaging.
* Participation in another clinical trial.
* Prior and/or current treatment with experimental immunotherapeutics including IVIG or vaccines for AD.
* Prior and/or current treatment with immunosuppressive drugs
* History and/or presence of autoimmune disease.

Other Exclusion Criteria apply.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2008-02; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Tolerability | 1 year

SECONDARY OUTCOMES:
Immunological and clinical efficacy (evaluated in explorative manner) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Margot Schmitz, Univ. Doz. Dr., Principal Investigator — Ordination Univ. Doz. Dr. Margot Schmitz
Locations (1):
- Ordination Univ. Doz. Dr. Margot Schmitz, Vienna, Austria